CLINICAL TRIAL: NCT02654561
Title: Phase 3 Study of the Efficacy and Safety of Unfractionated Heparin in Patients With Severe Sepsis/Septic Shock With Suspected DIC
Brief Title: Efficacy and Safety of Unfractionated Heparin on Severe Sepsis With Suspected Disseminated Intravascular Coagulation
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University, China (Other)
Collaborators: West China Hospital (Other); Zhongda Hospital (Other); The First Affiliated Hospital of Dalian Medical University (Other); Shengjing Hospital (Other); The First Hospital of Jilin University (Other); Qilu Hospital of Shandong University (Other); The Second Affiliated Hospital of Kunming Medical University (Other); The First Hospital of Qinhuangdao (Other Government); The Second Affiliated Hospital of Dalian Medical University (Other); First Affiliated Hospital of Harbin Medical University (Other); Peking University People's Hospital (Other); The People's Hospital of Liaoning Province (Other); Fourth People's Hospital of Shenyang (Other); Beijing Tsinghua Changgeng Hospital (Other); First Affiliated Hospital of Kunming Medical University (Other); The Affiliated Hospital of Qingdao University (Other); Beijing Friendship Hospital (Other); General Hospital of Ningxia Medical University (Other); The First Affiliated Hospital of Nanchang University (Other)
Responsible Party: Principal Investigator, Xiaochun Ma,MD, MD,PhD, China Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LNCCC-B01-2014
Record Dates: First submitted 2015-08-25; First posted 2016-01-13 (Estimated); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Sepsis; Disseminated Intravascular Coagulation
Keywords: Severe sepsis; Disseminated intravascular coagulation; Unfractionated heparin
MeSH Terms: conditions — Sepsis; Disseminated Intravascular Coagulation | interventions — Heparin; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Saline (Placebo Comparator)
  Interventions: Drug: Saline
- Heparin (Experimental): If severe sepsis with suspected DIC is diagnosed, the Heparin sodium(2ml:12500 units) will be administered intravenously continuously for 24 hours. The course of treatment will last 7 days or until the death or discharge.
  Interventions: Drug: Heparin Sodium; Drug: Saline

INTERVENTIONS:
Drug: Heparin Sodium — A bottle solution of Heparin Sodium(2ml:12500IU) is added to 50ml saline and administered i.v. continuously for 24 hours, which last 7 days or until the death or discharge. The same amount of 0.9% saline as the heparin group will be administered in the placebo group.
  Other Names: Unfractionated heparin
  Arms: Heparin
Drug: Saline — For all the severe sepsis or septic shock patients, normal saline will be administered for fluid resuscitation according to the Guideline of Survival Sepsis Campaign.
  Other Names: Normal saline

SUMMARY:
The primary objective of this study is to estimate the efficacy of unfractionated heparin(UFH) on ICU mortality in severe sepsis with suspected DIC.The Second objective is to estimate the effect of UFH on 28-day mortality,and the change of the Japanese Association for Acute Medicine(JAAM) score and SOFA score. The third one is to evaluate the safety of UFH in severe sepsis patients with suspected DIC.

DETAILED DESCRIPTION:
During the study, the whole process of data validation and registry procedures will be implemented by the Principal Investigator of the study, and monitored by the Ethics Committee of the First Affiliated Hospital of China Medical University.There are 2 research supervisors(2 ICU doctors) to assess the accuracy, completeness and representativeness of registry data, and to report the study process and research results to Principal Investigator.Investigators have also edited a data dictionary including each variable used by the registry and normal ranges of all detection indexes. The standard operating procedures have been formulated to address the registry and data analysis. The feasibility and significance have been assessed carefully and funded by the Health and Family Planning Commission of Liaoning Province(No.LNCC-B01-2014).The sample size is 600 participants through statistic calculation. The plan for missing data and statistical analysis will be implemented by specialized statisticians of China Medical University.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of severe sepsis or/and septic shock
* suspected DIC:the score of Platelets plus International Normalized Ratio in the JAAM criteria is equal or more than 3 scores

Exclusion Criteria:

* consent declined
* pregnant or breastfeeding
* the length during ICU is less than 24 hours
* with other types of shock
* have bleeding or high risk for bleeding
* have an indication for therapeutic anticoagulation
* have a known or suspected adverse reaction to UFH including HIT
* are currently enrolled in another trial
* known or suspected cirrhosis or other severe hepatic diseases
* terminal illness with a life expectancy of less than 28 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2018-04-12 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
ICU mortality | during ICU stay (up to day 28)
  The mortality during ICU stay

SECONDARY OUTCOMES:
28-day all-cause mortality | after 28 days of enrollment of all the cases
  The all-cause mortality at day 28 after enrollment
the incidence of major bleeding | during ICU stay (up to day 28)
  "Major bleeding" is defined as intracranial bleeding, life-threatening bleeding, or need red blood cell suspension more than 3 units every 24 hours,and last for 2 days

OTHER OUTCOMES:
Change in SOFA scores | during the intervention period (up to day 7 after enrollment)
  The difference of SOFA scores between day 7 and day 1 upon enrollment
Change in JAAM and ISTH scores | during the intervention period (up to day 7 upon enrollment)
  The difference of JAAM and ISTH scores between day7 and day1 upon enrollment

CONTACTS AND LOCATIONS:
Locations (17):
- China (17):
  - The fist Affiliated Hospital Harbin Medical University, Haerbin, Heilongjiang
  - Xiangya Third Hospital of Central South University, Changsha, Hunan
  - Zhongda Hospital, Nanjing, Jiangsu
  - First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - Second Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - second Affiliated Hospital of china Medical University, Shenyang, Liaoning
  - Shenyang Fourth People's Hospital, Shenyang, Liaoning
  - Qilu Hospital of Shandong University（qingdao）, Qingdao, Shandong
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - the Second Affiliated Hospital of Kunming University, Kunming, Yunnan
  - Beijing Friendship Hospital ， Capital Medical University, Beijing
  - Changgeng Hospital of Tsinghua University, Beijing
  - People's Hospital of Peking University, Beijing
  - First Affiliated Hospital of Jilin Medical University, Jilin
  - Qinhuangdao First Hospital, Qinhuangdao
  - Liaoning Provincial People's Hospital, Shenyang

REFERENCES:
- [Background] Zhang XJ, Ma XC. [Therapeutic effects of early administration of low-dose heparin in patients with severe sepsis]. Zhonghua Wai Ke Za Zhi. 2006 Sep 1;44(17):1209-11. Chinese. PMID 17147870
- [Background] Zhao C, Zhang ZD, Zhang XJ, Li X, Zhu R, Ma XC. [Evaluation of clinical effects on low-dose heparin therapy for sepsis]. Zhonghua Nei Ke Za Zhi. 2009 Jul;48(7):566-9. Chinese. PMID 19957797
- [Background] Jaimes F, De La Rosa G, Morales C, Fortich F, Arango C, Aguirre D, Munoz A. Unfractioned heparin for treatment of sepsis: A randomized clinical trial (The HETRASE Study). Crit Care Med. 2009 Apr;37(4):1185-96. doi: 10.1097/CCM.0b013e31819c06bc. PMID 19242322
- [Background] Liu XL, Wang XZ, Liu XX, Hao D, Jaladat Y, Lu F, Sun T, Lv CJ. Low-dose heparin as treatment for early disseminated intravascular coagulation during sepsis: A prospective clinical study. Exp Ther Med. 2014 Mar;7(3):604-608. doi: 10.3892/etm.2013.1466. Epub 2013 Dec 31. PMID 24520253
- [Background] Barkun J, Christou NV; CAGS Evidence Based Reviews in Surgery Group. Canadian Association of General Surgeons Evidence Based Reviews in Surgery. 8. Efficacy and safety of recombinant human activated protein C for severe sepsis. Can J Surg. 2003 Dec;46(6):468-70. No abstract available. PMID 14680357
- [Derived] Sun Y, Ding R, Sun H, Liang Y, Ma X. Efficacy and safety of heparin for sepsis-induced disseminated intravascular coagulation (HepSIC): study protocol for a multicenter randomized controlled trial. Trials. 2024 Jan 2;25(1):4. doi: 10.1186/s13063-023-07853-5. PMID 38167115